CLINICAL TRIAL: NCT03708718
Title: A Phase II Randomised Study of Oral Prednisolone in Early Diffuse Cutaneous Systemic Sclerosis (Initially Double-blind, Then Switched to Open-label Because of Covid-19)
Brief Title: Prednisolone in Early Diffuse Systemic Sclerosis
Acronym: PRedSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Ariane herrick (Other)
Collaborators: Versus Arthritis (Other)
Responsible Party: Sponsor-Investigator, Prof. Ariane herrick, Professor of Rheumatology, University of Manchester
Organization: University of Manchester (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 119220
Record Dates: First submitted 2018-10-08; First posted 2018-10-17 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Systemic Sclerosis
Keywords: Diffuse cutaneous systemic sclerosis (dcSSc); Prednisolone; Randomised Controlled Trial; Disability; Pain; Fatigue
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Pain; Fatigue | interventions — Prednisolone

STUDY DESIGN:
Intervention Model Description: Patients are allocated to received either prednisolone or matched placebo for the duration of the trial. The allocation is randomised 1:1.
  From August 2020: Under the open-label design, patients are allocated to receive prednisolone or no additional treatment. The randomisation allocation is 1:1.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind. The trial management team are blind to treatment allocation for the duration of the trial. The site research teams and patients are blind to treatment until code-break. At this point the on-site team and patient are unblind to allocation for continuing care. The site pharmacy personnel, PRedSS trial monitor and supervising statistician are unblind throughout.
  From August 2020: Open-Label - The patient, site research team and site pharmacy are unblind. The trial management team are unblind for patients recruited from August 2020 onwards but remain blind to patients randomised to trial under the double-blind design. The trial monitor and trial statistician continue to be unblind for all patients randomised to trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisolone (Active Comparator): Prednisolone 5mg enteric-coated tablets, over-encapsulated in a hard gelatine capsule and filled with lactose BP. The prednisolone will be self-administered, orally with water before or after a meal once a day. Dosing will be continuous for a total of 6 months.
  The total dose prescribed will be equivalent to approximately 0.3mg/kg/day. The minimum dose prescribed will be 10mg per day (2 capsules) and a maximum of 30mg per day (6 capsules).
  From August 2020: The prednisolone is no longer over-encapsulated. Prednisolone 5mg enteric-coated tablets will be prescribed and taken as above.
  Interventions: Drug: Prednisolone 5 mg
- Placebo oral capsule; From August 2020 - 'no additional treatment' (Placebo Comparator): The placebo will be a hard gelatine capsule filled with lactose BP and identically matched to the prednisolone capsules. The placebo will be self-administered once a day, orally with water before or after a meal. Dosing will be continuous for a total of 6 months.
  From August 2020 - no placebo capsule will be administered.
  Interventions: Drug: Placebo oral capsule; From August 2020 'no additional treatment'

INTERVENTIONS:
Drug: Prednisolone 5 mg — 5mg prednisolone, once a day for 6 months
  Arms: Prednisolone
Drug: Placebo oral capsule; From August 2020 'no additional treatment' — Matched placebo capsule, once a day for 6 months; From August 2020 - no additional treatment above standard of care medication
  Arms: Placebo oral capsule; From August 2020 - 'no additional treatment'

SUMMARY:
This is a randomised placebo-controlled study of moderate dose prednisolone for 6 months in patients with early diffuse cutaneous systemic sclerosis (dcSSc). Seventy-two patients within 3 years of the onset of skin thickening will be recruited from 14 UK centres over 3 years. Co-primary end-points will be the Health Assessment Questionnaire Disability Index (HAQ-DI) and the modified Rodnan skin score (mRSS). Patients will be assessed 5 times: screening, baseline, 6 weeks, 3 and 6 months, with a code-break on exit from the study at 6 months.

Please note: From August 2020, the trial was re-started following halt due to Covid-19 as open-label. The placebo arm is the 'no treatment' arm and there is no longer a code-break at study exit.

DETAILED DESCRIPTION:
The study is a non-commercial phase II randomised, double-blind, placebo-controlled, multi-centre study to test moderate dose prednisolone versus placebo in patients with early diffuse cutaneous systemic sclerosis (dcSSc).

Our aim is to investigate whether treatment with the steroid prednisolone is beneficial in patients with early diffuse cutaneous systemic sclerosis (also termed "scleroderma"). This is a controversial subject. Although it is very possible that prednisolone can help relieve the severe pain, itching, and disability (due to contractures and musculoskeletal involvement) of early diffuse scleroderma, doctors are often reluctant to prescribe prednisolone because of possible side effects, particularly an increased risk of serious kidney problems. Our proposed trial, treating patients with either prednisolone or placebo therapy for 6 months, should provide clinicians with a long awaited answer to the important clinical question: Can prednisolone be used as a therapy in this group of patients?

The study, funded by Arthritis Research UK, aims to determine:

1. Is moderate dose prednisolone effective in reducing pain, disability and skin thickening in patients with early diffuse scleroderma?
2. Is moderate dose prednisolone a safe therapy in patients with early diffuse scleroderma (with particular reference to kidney function)?

If the answer to both is 'yes', then prednisolone therapy will be much more widely prescribed for this patient group.

The patient population will be selected from individuals with early dcSSc, as defined by skin involvement of less than 3 years, who are considered potentially able to benefit from this treatment. Following screening, to minimise bias, eligible patients will be randomised at the baseline visit to receive either daily moderate dose prednisolone (as determined by body weight) or a matched placebo. To further eliminate subjective and unrecognised bias both the research team and patients will be blind to the randomisation. A placebo control, as opposed to an active treatment control, will be administered. This is necessary as the study treatment is adjunctive to and not a substitute for any other therapies which may be prescribed, such as immunosuppressant therapies.

Patients will attend on 5 occasions (screen, baseline, 6 weeks, 3 and 6 months). All patients will be considered off-study at the end of the 6 month visit whereupon the treatment code will be broken. At each visit a number of measurements will be taken including functional ability, degree of skin involvement (skin score), mood and kidney function. This will allow us to determine whether 'active' (prednisolone) therapy is effective and free from serious side-effects.

Please note: from August 2020, due to Covid-19 the trial was re-designed and re-started following trial halt as open-label. A placebo is no longer required. The aims, primary outcome measures and number of visits remain unchanged. However, to further mitigate the ongoing impact of Covid-19, the screen and baseline assessments may now be conducted at the same visit. Remote visits can also be carried out at 6 weeks and 6 months, if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with dcSSc with skin involvement extending to the proximal limb and/or trunk.
2. Male or female age ≥ 18 years.
3. Skin involvement of less than 3 years defined by patient report or clinician opinion.
4. Patient is able and willing to follow the requirements of the study.
5. Fully written informed consent.

Exclusion Criteria:

1. Patients with significant uncontrolled Stage 1 Hypertension (clinic BP >140/90mmHg i.e. either >140mmHg OR >90mmHg). Patients with previous hypertension which is controlled (clinic BP <140/90mmHg) for at least 4 weeks are considered eligible.
2. Previous renal crisis or significant renal impairment (estimated Glomerular Filtration Rate (eGFR) < 40 ml/min).
3. Patients currently on steroid therapy, or previous steroid therapy within the last 4 weeks, with the exception of inhaled steroids for respiratory diseases.
4. Patients currently participating in another randomised controlled trial of an investigational agent or device, or previous participation within the last 30 days.
5. Patients currently receiving an immunosuppressant or biologic therapy the dose of which has changed in the last 4 weeks prior to the baseline visit, or is likely to change during the first 3 months of study treatment.
6. Patients with major myositis or inflammatory arthritis. Patients with low level myositis or inflammatory arthritis are eligible for inclusion (for example, in the case of myositis, a creatine kinase less than 4 times the upper limit of normal or myositis only demonstrable on magnetic resonance imaging).
7. Female patients who are pregnant at time of screening.
8. Female patients who are breastfeeding.
9. Patients with significant inflammatory bowel disease as judged by the investigator.
10. It is important that patients do not suddenly stop taking the study medication. Patients who do not fully understand this, will be excluded.
11. Patients who are unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Health Assessment Questionnaire Disability Index (HAQ-DI) | Baseline to 3 months
  The mean difference in HAQ-DI at 3 months
modified Rodnan Skin Score (mRSS) | Baseline to 3 months
  The difference in mRSS at 3 months

SECONDARY OUTCOMES:
Quality of life and functional ability - Assessed by Questionnaire | Baseline to 6 weeks and 6 months
  HAQ-DI
Pain and disability | Baseline to 6 weeks and 6 months
  Skin involvement as measured by the mRSS
Functional ability - Assessed by Questionnaire | Baseline to 6 weeks, 3 months and 6 months
  11-point Scleroderma Functional Index
Pain associated with itch - Assessed by Questionnaire | Baseline to 6 weeks, 3 months and 6 months
  Assessment of Pruritus
Hand function - Assessed by Questionnaire | Baseline to 6 weeks, 3 months and 6 months
  Cochin Hand Function
Fatigue - Assessed by Questionnaire | Baseline to 6 weeks, 3 months and 6 months
  Functional Assessment of Chronic Illness Therapy (FACIT)
Anxiety and depression - Assessed by questionnaire | Baseline to 6 weeks, 3 months and 6 months
  Hospital Anxiety and Depression Scale (HADS) . This questionnaire has 14 questions, each with 4 options designed to assess aspects of mental health
Health related quality of life - Assessed by Questionnaire | Baseline to 6 weeks, 3 months and 6 months
  Helplessness Questionnaire
Health related quality of life - Assessed by Questionnaire | Baseline to 6 weeks, 3 months and 6 months
  Short Form (36) Health Survey
Health related quality of Life - Assessed by Questionnaire | Baseline to 6 weeks, 3 months and 6 months
  EuroQol 5 Dimensions
Pain and disability | Baseline to 6 weeks, 3 months and 6 months
  Patient Global Assessment
Pain and disability | Baseline to 6 weeks, 3 months and 6 months
  Physician Global Assessment
Assessment of pain - Clinician assessment | Baseline to 6 weeks, 3 months and 6 months
  Digital Ulcer Count: The site and total number of ulcers on the hand are recorded by the patients clinician on a diagram of a hand
Assessment of pain - Clinician assessment | Baseline to 6 weeks, 3 months and 6 months
  Tender Friction Rubs - the total number of tendon friction rubs on 12 possible anatomical sites are recorded
Assessment of pain - Clinician assessment | Baseline to 6 weeks, 3 months and 6 months
  Joint Count: The number of tender or swollen joints are assessed from 14 anatomical sites (both left and right side) and recorded out of a total of 28 (14 sites, left and right side) tender joints and 28 swollen joints
Pain and disability - Assessed by Questionnaire | Baseline to 6 weeks, 3 months and 6 months
  Assessment of Arthritis Index
Pain and disability | Baseline to 6 weeks, 3 months and 6 months
  Assessment in percentage change of mRSS

CONTACTS AND LOCATIONS:
Overall Officials: Professor Ariane Herrick, Principal Investigator — University of Manchester
Locations (14):
- United Kingdom (14):
  - Aberdeen Royal Infirmary - NHS Grampian, Aberdeen, Aberdeenshire
  - Addenbrooke's Hospital - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - Salford Royal NHS Foundation Trust, Salford, Greater Manchester
  - Glasgow Royal Infirmary -, Glasgow, Lanarkshire
  - Aintree University Hospitals NHS Foundation Trust, Liverpool, Merseyside
  - Queen's Medical Centre - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - Royal National Hospital For Rheumatic Diseases - Royal United Hospitals Bath NHS Foundation Trust, Bath, Somerset
  - Royal Hallamshire Hospital - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire
  - Freeman Hospital - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne and Wear
  - The Dudley Group NHS Foundation Trust, Dudley, West Midlands
  - Leeds Institute of Rheumatic and Musculoskeletal Medicine, Leeds, West Yorkshire
  - Southmead Hospital Bristol - North Bristol NHS Trust, Bristol
  - Ninewells Hospital and Medical School - NHS Tayside, Dundee
  - Royal Free London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared with collaborating centres. It is undecided if this information will be shared with researchers unconnected with the trial.

REFERENCES:
- [Derived] Griffiths-Jones DJ, Garcia YS, Ryder WD, Pauling JD, Hall F, Lanyon P, Bhat S, Douglas K, Gunawardena H, Akil M, Anderson M, Griffiths B, Del Galdo F, Youssef H, Madhok R, Arthurs B, Buch M, Fligelstone K, Zubair M, Mason JC, Denton CP, Herrick AL. A Phase II randomized controlled trial of oral prednisolone in early diffuse cutaneous systemic sclerosis (PRedSS). Rheumatology (Oxford). 2023 Sep 1;62(9):3133-3138. doi: 10.1093/rheumatology/kead012. PMID 36637209